CLINICAL TRIAL: NCT00438724
Title: A Randomized Control Trial of an Intervention for Couples Coping With Alzheimer's Disease
Brief Title: Couples Coping With Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alzheimer's Association (Other)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IA0103; ZEN-04-1011
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Aging; Alzheimer Disease; Dementia
Keywords: Caregivers; Caregiving; Spousal relationships; cognition disorders; therapy; mental health; psychosocial
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognition Disorders; Psychological Well-Being | interventions — Counseling; Palliative Care

INTERVENTIONS:
Behavioral: Information, counseling and support

SUMMARY:
The purpose of this study is to test the efficacy of a new couples counseling intervention for people recently diagnosed with early Alzheimer's disease and their spouses. The study hypothesis is that counseling the couple shortly after the diagnosis, and while the functional impact of the illness is still relatively mild, will have a significant impact on their ability to provide support for each other.

DETAILED DESCRIPTION:
The majority of people with Alzheimer's disease (AD) live at home with their spouses. AD erodes the ability of each member of the couple to support each other. Moreover, couples may be unaccustomed to seeking or accepting emotional and practical support from family members or formal resources. Even though AD can have a major negative impact on each member of the couple and on their relationship, their needs have generally been addressed separately, often without sufficient appreciation for the importance of their ongoing relationship. Previous studies suggest that by improving support for both members of the couple, the intervention will have a positive effect on mental health outcomes such as depression and help keep the person with AD at home rather than in a long-term care facility.

One hundred couples will be randomly assigned either to an immediate treatment group or a wait-list control group which will receive treatment four months after enrollment. Participants will receive a formal baseline assessment, consisting of a structured set of questionnaires to assess dyadic (couple) adjustment, social support, depression and anxiety as well as goals for counseling. There will be two follow-up assessments, 2 and 4 months after baseline using the same instruments. All participants will be able to call a counselor for the duration of the study to obtain resource and referral information or in the event of a crisis. The treatment will consist of 6 sessions of couples counseling within a 2-month period. The focus will be on helping each member of the couple to express feelings, needs and issues that have emerged between them as a result of the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Couples, in which one partner has been diagnosed with AD and is in the mild stage of the disease
* Ages 21 to 90

Exclusion Criteria:

* Severe psychological or physical illness
* Unwillingness to participate in all aspects of the study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-11; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Changes in dyadic (couple) adjustment
depression

SECONDARY OUTCOMES:
Level of anxiety
satisfaction with social support

CONTACTS AND LOCATIONS:
Overall Officials: Mary S. Mittelman, DrPH, Principal Investigator — NYU School of Medicine
Locations (1):
- Aging and Dementia Research Center, Silberstein Institute, NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Morrissey MV. Rethinking the benefits of an adapted version of 'Alzheimer Cafe' for individuals with Alzheimer's and their partners. Int J Psychiatr Nurs Res. 2006 Sep;12(1):1393-401. PMID 17016901
- [Background] Robinson L, Clare L, Evans K. Making sense of dementia and adjusting to loss: psychological reactions to a diagnosis of dementia in couples. Aging Ment Health. 2005 Jul;9(4):337-47. doi: 10.1080/13607860500114555. PMID 16019290
- [Background] Gallagher-Thompson D, Dal Canto PG, Jacob T, Thompson LW. A comparison of marital interaction patterns between couples in which the husband does or does not have Alzheimer's disease. J Gerontol B Psychol Sci Soc Sci. 2001 May;56(3):S140-50. doi: 10.1093/geronb/56.3.s140. PMID 11316839
- [Background] Auclair U, Epstein C, Mittelman M. Couples Counseling in Alzheimer's Disease: Additional Clinical Findings from a Novel Intervention Study. Clin Gerontol. 2009 Apr 1;32(2):130-146. doi: 10.1080/07317110802676809. PMID 19865591